CLINICAL TRIAL: NCT01464164
Title: Phase I/II, Open-Label Study to Determine Safety and Efficacy of Sotatercept (ACE-011) in Adults With Red Blood Cell Transfusion- Dependent Diamond Blackfan Anemia
Brief Title: Safety and Efficacy Study of Sotatercept in Adults With Transfusion Dependent Diamond Blackfan Anemia
Acronym: ACE-011-DBA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Supporter terminated the study due to no active patients (secondary to travel restrictions due to COVID).
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Adrianna Vlachos, MD, Principal Investigator, Northwell Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-02-199 - 06A
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Diamond Blackfan Anemia
Keywords: Diamond Blackfan anemia; DBA; Blackfan Diamond anemia; Congenital pure red cell aplasia; Aase-Smith II Syndrome; Aase Syndrome; Anemia, Congenital Pure Red Cell; Aplasia, Congenital Pure Red Cell; BDA; Congenital Hypoplastic Anemia; Erythrogenesis Imperfecta; Hypoplastic Congenital Anemia; Inherited Erythroblastopenia; pure red cell aplasia; bone marrow failure syndrome
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Anemia, Hypoplastic, Congenital; Aase Smith syndrome 2; Red-Cell Aplasia, Pure; Bone Marrow Failure Disorders | interventions — ACE-011; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotatercept (Experimental): Sotatercept to be given as a subcutaneous injection once a month for 4 consecutive months, using a dose escalation scale among 3 cohorts. *Protocol Amendment: Two additional cohorts will be given Sotatercept 0.75mg/kg and 1 mg/kg as a subcutaneous injection once every 3 weeks.
  Interventions: Drug: Sotatercept
- Sotatercept with prednisone boost (Experimental): Protocol Amendment: Two additional cohorts will be given Sotatercept 0.75mg/kg and 1 mg/kg as a subcutaneous injection once every 3 weeks along with a prednisone boost of 1 mg/kg daily for 3 weeks (max of 60 mg).
  Interventions: Drug: Sotatercept with prednisone boost

INTERVENTIONS:
Drug: Sotatercept — Cohort 4a: 3 patients on Sotatercept 0.75 mg/kg every 3 weeks. If the patients have no untoward events in the Patients in Dose Level 4 by the end of 3 of the 6 doses, then additional patients (Dose Level 5) will be enrolled at the next dose level:
  Cohort 5a: 3 patients on Sotatercept 1 mg/kg every 3 weeks
  Other Names: ACE-011
  Arms: Sotatercept
Drug: Sotatercept with prednisone boost — Cohort 4b: 3 patients on Sotatercept 0.75 mg/kg every 3 weeks with a three week prednisone boost of 1 mg/kg/day (max 60 mg). If the patients have no untoward events in the Patients in Dose Level 4 by the end of 3 of the 6 doses, then additional patients (Dose Level 5) will be enrolled at the next dose level:
  Cohort 5b: 3 patients on Sotatercept 1 mg/kg every 3 weeks with a 3 week prednisone boost of 1 mg/kg/day (max 60 mg).
  Other Names: ACE-011 and Prednisone
  Arms: Sotatercept with prednisone boost

SUMMARY:
The purpose of this study is to determine the safety and dosing of drug Sotatercept, as a subcutaneous injection, to stimulate production of red blood cell production. To be given every 28 days for up to four doses.

DETAILED DESCRIPTION:
This study is for adult patients with Diamond Blackfan Anemia who are currently being transfused every 3- 4 weeks.

The drug will be given as a subcutaneous injection within one of three dose levels. The first dose level (0.1 mg/kg) will include 3 subjects who will receive the same dose of the drug monthly for a total of 4 doses, as long as there are no dose- limiting toxicities (DLTs). A Dose limiting toxicity is defined as inability to deliver the scheduled doses because of toxicity >/= Grade 3, according to NCI Toxicity Grading Scale.

Once all 3 subjects have received and tolerated the low dose level, the next level will open (0.3 mg/kg)to 3 new subjects. Subjects will be monitored closely for response and side effects.

If more than 2 subjects have a dose limiting toxicity in the first dose level, then dose level -1 (0.05 mg/kg)will open, enrolling 3 more subjects. If more than 2 subjects at dose level -1, have dose limiting toxicities, the study will be discontinued. If there are no additional dose limiting toxicities, dose level -1 will be the maximum tolerated dose.

There are a total of 3 dose levels, not including dose level -1. Once the maximum tolerated dose has been reached, up to a total of 10 additional subjects will be enrolled.

Protocol Amendment: The protocol has been amended to include an additional enrollment of 20 subjects with two additional dose levels of Sotatercept (0.075 mg/kg and 0.100 mg/kg ) to be given with or without a prednisone boost.

Efficacy will be measured by response. A complete response will be determined if the subject no longer requires transfusion, while on study drug. A partial response will be measured by a reduction by 50% in need for transfusion.

Treatment modifications will be made based on evidence of side effects. Dose- escalation will be performed only if no side effects are reported and no efficacy is evidenced. Treatment will be stopped if hemoglobin is >12 gm/dl and/ or any >/+ grade 3 adverse event is related to sotatercept.

Study assessments will include:

* Physical exam (height, weight, vital signs and blood pressure)at screening, day 1 of each cycle and monthly for 3 months of follow up period as well as at study discontinuation.
* Additional blood pressure monitoring at day 1 of each cycle and weekly there after through cycle 4, monthly in follow up period and at study discontinuation.
* Karnofsky performance status at screening, day 1 of cycle 2 and day 1 of monthly follow up period for 3 months and study discontinuation.
* CBC reticulocyte count and ANC will be collected at day 1 of each cycle and weekly there after through cycle 4, monthly in follow up period and at study discontinuation.
* Blood chemistry, liver and kidney function will be assessed at screening, day 1 and 15 of cycle 1, day 1 of cycle 2, 3, 4 month 1 in follow up and at study discontinuation.
* Blood for iron status (serum iron, transferrin and %, ferritin) will be collected during the screening period, and at month 1 of the follow-up period as well as study discontinuation.
* Folate and B12 levels will be assessed during the screening period at day 1 of cycle 3 and again at study discontinuation.
* Urinalysis (creatinine, protein),at screening, day 15 of cycle 1, day 1 of cycles 2, 3, and 4 monthly during follow-up and at study discontinuation.
* Serum erythropoietin at screening, day 15 of cycle 1, day 1 of cycle 3, monthly during follow-up and at study discontinuation.
* FSH & LH (everyone), DHEA & testosterone (males only), estrogen & estradiol (females only)at screening, day 1 of cycles 2, 3, and 4, monthly during follow- up period and at study discontinuation.
* EKG & ECHO at screening, day 1 of cycle 3 first month of follow-up period and at study discontinuation
* Dexa Scan at screening, day 1 of monthly follow-up period and at study discontinuation
* Transfusion assessment at screening, day 1, 8, 15 and 22 of cycle 1, day 1 and 15 of cycles 2, 3, and 4, monthly during follow-up period and at study discontinuation.
* Response assessment at day 8, 15, 22 of cycle 1, day 1 and 15 of cycles2, 3, and 4, monthly for 3 months during follow-up period and at study discontinuation
* Adverse events, concomitant therapies to be assessed at day 1, 8, 15, and 22 of cycle 1, day 1 and 15 of cycles 2, 3, and 4, monthly during follow-up period and at study discontinuation
* Drug administration day 1 of cycles 1, 2, 3, and 4.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age
* DBA diagnosed
* RBC transfusion- dependence (defined as >/= 10 cc/kg of RBC per 28 days average)
* Karnofsky performance scale >/= 70
* Females of childbearing potential are to use birth control during study participation and for 112 days following the last dose of sotatercept
* Males must agree to use a latex condom during any sexual contact with females of childbearing potential while participating in the study and for 112 days following the last dose of sotatercept
* Agreement to adhere to the study visit schedule, understand and comply with all protocol requirements
* Understand and sign a written informed consent

Exclusion Criteria:

* Creatinine clearance < 30 ml/min
* SGOT > 3x upper limit of normal, SGPT > 3x upper limit normal, or bilirubin >3x upper limit normal
* Heart disease (NY Heart Association classification of >/= 3
* History of hypertension
* Subjects currently responsive to corticosteroids for treatment of Diamond Blackfan anemia
* Treatment with another investigational drug or device <56 days pre-study entry
* Pregnant or lactating females
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrianna Vlachos, MD, Principal Investigator — Northwell Health/Feinstein Institute for Medical Research
Locations (1):
- North Shore- LIJ campus of The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abkowitz JL, Schaison G, Boulad F, Brown DL, Buchanan GR, Johnson CA, Murray JC, Sabo KM. Response of Diamond-Blackfan anemia to metoclopramide: evidence for a role for prolactin in erythropoiesis. Blood. 2002 Oct 15;100(8):2687-91. doi: 10.1182/blood.V100.8.2687. PMID 12351372
- [Background] Diamond LK, Wang WC, Alter BP. Congenital hypoplastic anemia. Adv Pediatr. 1976;22:349-78. PMID 773132
- [Background] Ball SE, McGuckin CP, Jenkins G, Gordon-Smith EC. Diamond-Blackfan anaemia in the U.K.: analysis of 80 cases from a 20-year birth cohort. Br J Haematol. 1996 Sep;94(4):645-53. doi: 10.1046/j.1365-2141.1996.d01-1839.x. PMID 8826887
- [Background] Bastion Y, Bordigoni P, Debre M, Girault D, Leblanc T, Tchernia G, Ball S, McGuckin C, Gordon-Smith EC, Bekassy A, et al. Sustained response after recombinant interleukin-3 in diamond blackfan anemia. Blood. 1994 Jan 15;83(2):617-8. No abstract available. PMID 8286756
- [Background] Cmejla R, Cmejlova J, Handrkova H, Petrak J, Pospisilova D. Ribosomal protein S17 gene (RPS17) is mutated in Diamond-Blackfan anemia. Hum Mutat. 2007 Dec;28(12):1178-82. doi: 10.1002/humu.20608. PMID 17647292
- [Background] Da Costa L, Moniz H, Simansour M, Tchernia G, Mohandas N, Leblanc T. Diamond-Blackfan anemia, ribosome and erythropoiesis. Transfus Clin Biol. 2010 Sep;17(3):112-9. doi: 10.1016/j.tracli.2010.06.001. Epub 2010 Jul 23. PMID 20655265
- [Background] Doherty L, Sheen MR, Vlachos A, Choesmel V, O'Donohue MF, Clinton C, Schneider HE, Sieff CA, Newburger PE, Ball SE, Niewiadomska E, Matysiak M, Glader B, Arceci RJ, Farrar JE, Atsidaftos E, Lipton JM, Gleizes PE, Gazda HT. Ribosomal protein genes RPS10 and RPS26 are commonly mutated in Diamond-Blackfan anemia. Am J Hum Genet. 2010 Feb 12;86(2):222-8. doi: 10.1016/j.ajhg.2009.12.015. Epub 2010 Jan 28. PMID 20116044
- [Background] Draptchinskaia N, Gustavsson P, Andersson B, Pettersson M, Willig TN, Dianzani I, Ball S, Tchernia G, Klar J, Matsson H, Tentler D, Mohandas N, Carlsson B, Dahl N. The gene encoding ribosomal protein S19 is mutated in Diamond-Blackfan anaemia. Nat Genet. 1999 Feb;21(2):169-75. doi: 10.1038/5951. PMID 9988267
- [Background] Farrar JE, Nater M, Caywood E, McDevitt MA, Kowalski J, Takemoto CM, Talbot CC Jr, Meltzer P, Esposito D, Beggs AH, Schneider HE, Grabowska A, Ball SE, Niewiadomska E, Sieff CA, Vlachos A, Atsidaftos E, Ellis SR, Lipton JM, Gazda HT, Arceci RJ. Abnormalities of the large ribosomal subunit protein, Rpl35a, in Diamond-Blackfan anemia. Blood. 2008 Sep 1;112(5):1582-92. doi: 10.1182/blood-2008-02-140012. Epub 2008 Jun 5. PMID 18535205
- [Background] Gale RP, Barosi G, Barbui T, Cervantes F, Dohner K, Dupriez B, Gupta V, Harrison C, Hoffman R, Kiladjian JJ, Mesa R, Mc Mullin MF, Passamonti F, Ribrag V, Roboz G, Saglio G, Vannucchi A, Verstovsek S. What are RBC-transfusion-dependence and -independence? Leuk Res. 2011 Jan;35(1):8-11. doi: 10.1016/j.leukres.2010.07.015. Epub 2010 Aug 7. PMID 20692036
- [Background] Gazda HT, Grabowska A, Merida-Long LB, Latawiec E, Schneider HE, Lipton JM, Vlachos A, Atsidaftos E, Ball SE, Orfali KA, Niewiadomska E, Da Costa L, Tchernia G, Niemeyer C, Meerpohl JJ, Stahl J, Schratt G, Glader B, Backer K, Wong C, Nathan DG, Beggs AH, Sieff CA. Ribosomal protein S24 gene is mutated in Diamond-Blackfan anemia. Am J Hum Genet. 2006 Dec;79(6):1110-8. doi: 10.1086/510020. Epub 2006 Nov 2. PMID 17186470
- [Background] Gazda HT, Sheen MR, Vlachos A, Choesmel V, O'Donohue MF, Schneider H, Darras N, Hasman C, Sieff CA, Newburger PE, Ball SE, Niewiadomska E, Matysiak M, Zaucha JM, Glader B, Niemeyer C, Meerpohl JJ, Atsidaftos E, Lipton JM, Gleizes PE, Beggs AH. Ribosomal protein L5 and L11 mutations are associated with cleft palate and abnormal thumbs in Diamond-Blackfan anemia patients. Am J Hum Genet. 2008 Dec;83(6):769-80. doi: 10.1016/j.ajhg.2008.11.004. PMID 19061985
- [Background] Glader BE, Backer K, Diamond LK. Elevated erythrocyte adenosine deaminase activity in congenital hypoplastic anemia. N Engl J Med. 1983 Dec 15;309(24):1486-90. doi: 10.1056/NEJM198312153092404. PMID 6646173
- [Background] Gustavsson P, Skeppner G, Johansson B, Berg T, Gordon L, Kreuger A, Dahl N. Diamond-Blackfan anaemia in a girl with a de novo balanced reciprocal X;19 translocation. J Med Genet. 1997 Sep;34(9):779-82. doi: 10.1136/jmg.34.9.779. PMID 9321770
- [Background] Leblanc TM, Da Costa L, Marie I, Demolis P, Tchernia G. Metoclopramide treatment in DBA patients: no complete response in a French prospective study. Blood. 2007 Mar 1;109(5):2266-7. doi: 10.1182/blood-2006-08-039545. No abstract available. PMID 17312003
- [Background] Lipton JM, Atsidaftos E, Zyskind I, Vlachos A. Improving clinical care and elucidating the pathophysiology of Diamond Blackfan anemia: an update from the Diamond Blackfan Anemia Registry. Pediatr Blood Cancer. 2006 May 1;46(5):558-64. doi: 10.1002/pbc.20642. PMID 16317735
- [Background] Lipton JM, Kudisch M, Gross R, Nathan DG. Defective erythroid progenitor differentiation system in congenital hypoplastic (Diamond-Blackfan) anemia. Blood. 1986 Apr;67(4):962-8. PMID 3955239
- [Background] Liu JM, Ellis SR. Ribosomes and marrow failure: coincidental association or molecular paradigm? Blood. 2006 Jun 15;107(12):4583-8. doi: 10.1182/blood-2005-12-4831. Epub 2006 Feb 28. PMID 16507776
- [Background] Murata M, Onomichi K, Eto Y, Shibai H, Muramatsu M. Expression of erythroid differentiation factor (EDF) in Chinese hamster ovary cells. Biochem Biophys Res Commun. 1988 Feb 29;151(1):230-5. doi: 10.1016/0006-291x(88)90583-9. PMID 3348775
- [Background] Narla A, Vlachos A, Nathan DG. Diamond Blackfan anemia treatment: past, present, and future. Semin Hematol. 2011 Apr;48(2):117-23. doi: 10.1053/j.seminhematol.2011.01.004. PMID 21435508
- [Background] Nishiura H, Tanase S, Shibuya Y, Futa N, Sakamoto T, Higginbottom A, Monk P, Zwirner J, Yamamoto T. S19 ribosomal protein dimer augments metal-induced apoptosis in a mouse fibroblastic cell line by ligation of the C5a receptor. J Cell Biochem. 2005 Feb 15;94(3):540-53. doi: 10.1002/jcb.20318. PMID 15543555
- [Background] Ohene-Abuakwa Y, Orfali KA, Marius C, Ball SE. Two-phase culture in Diamond Blackfan anemia: localization of erythroid defect. Blood. 2005 Jan 15;105(2):838-46. doi: 10.1182/blood-2004-03-1016. Epub 2004 Jul 6. PMID 15238419
- [Background] Perrien DS, Akel NS, Edwards PK, Carver AA, Bendre MS, Swain FL, Skinner RA, Hogue WR, Nicks KM, Pierson TM, Suva LJ, Gaddy D. Inhibin A is an endocrine stimulator of bone mass and strength. Endocrinology. 2007 Apr;148(4):1654-65. doi: 10.1210/en.2006-0848. Epub 2006 Dec 28. PMID 17194739
- [Background] Quarello P, Garelli E, Carando A, Brusco A, Calabrese R, Dufour C, Longoni D, Misuraca A, Vinti L, Aspesi A, Biondini L, Loreni F, Dianzani I, Ramenghi U. Diamond-Blackfan anemia: genotype-phenotype correlations in Italian patients with RPL5 and RPL11 mutations. Haematologica. 2010 Feb;95(2):206-13. doi: 10.3324/haematol.2009.011783. Epub 2009 Sep 22. PMID 19773262
- [Background] Rivier J, Spiess J, McClintock R, Vaughan J, Vale W. Purification and partial characterization of inhibin from porcine follicular fluid. Biochem Biophys Res Commun. 1985 Nov 27;133(1):120-7. doi: 10.1016/0006-291x(85)91849-2. PMID 4074357
- [Background] Ruckle J, Jacobs M, Kramer W, Pearsall AE, Kumar R, Underwood KW, Seehra J, Yang Y, Condon CH, Sherman ML. Single-dose, randomized, double-blind, placebo-controlled study of ACE-011 (ActRIIA-IgG1) in postmenopausal women. J Bone Miner Res. 2009 Apr;24(4):744-52. doi: 10.1359/jbmr.081208. PMID 19049340
- [Background] Vlachos A, Ball S, Dahl N, Alter BP, Sheth S, Ramenghi U, Meerpohl J, Karlsson S, Liu JM, Leblanc T, Paley C, Kang EM, Leder EJ, Atsidaftos E, Shimamura A, Bessler M, Glader B, Lipton JM; Participants of Sixth Annual Daniella Maria Arturi International Consensus Conference. Diagnosing and treating Diamond Blackfan anaemia: results of an international clinical consensus conference. Br J Haematol. 2008 Sep;142(6):859-76. doi: 10.1111/j.1365-2141.2008.07269.x. Epub 2008 Jul 30. PMID 18671700
- [Background] Vlachos A, Muir E. How I treat Diamond-Blackfan anemia. Blood. 2010 Nov 11;116(19):3715-23. doi: 10.1182/blood-2010-02-251090. Epub 2010 Jul 22. PMID 20651069
- [Background] Vlachos A, Federman N, Reyes-Haley C, Abramson J, Lipton JM. Hematopoietic stem cell transplantation for Diamond Blackfan anemia: a report from the Diamond Blackfan Anemia Registry. Bone Marrow Transplant. 2001 Feb;27(4):381-6. doi: 10.1038/sj.bmt.1702784. PMID 11313667
- [Background] Vlachos A, Klein GW, Lipton JM. The Diamond Blackfan Anemia Registry: tool for investigating the epidemiology and biology of Diamond-Blackfan anemia. J Pediatr Hematol Oncol. 2001 Aug-Sep;23(6):377-82. doi: 10.1097/00043426-200108000-00015. PMID 11563775

RESULTS

PARTICIPANT FLOW:
Groups:
- Sotatercept Cohort 1: Cohort 1: Sotatercept 0.1 mg/kg given as a subcutaneous injection once every 4 weeks - to be completed in 3 patients without untoward events
- Sotatercept Cohort 2: Cohort 2: Sotatercept 0.3 mg/kg given as a subcutaneous injection once every 4 weeks - to be completed in 3 patients without untoward events
- Sotatercept Cohort 3: Cohort 3: Sotatercept 0.5 mg/kg given as a subcutaneous injection once every 4 weeks - to be completed in 3 patients without untoward events
- Sotatercept With Prednisone Boost Cohort 4a: Cohort 4a: Sotatercept 0.75 mg/kg given as a subcutaneous injection every 3 weeks with a three week prednisone boost of 1 mg/kg/day (max 60 mg) - to be completed in 3 patients without untoward events
- Sotatercept Cohort 4b: Cohort 4b: Sotatercept 0.75 mg/kg given as a subcutaneous injection every 3 weeks - to be completed in 3 patients without untoward events
- Sotatercept With Prednisone Boost Cohort 5a: Cohort 5a: Sotatercept 1 mg/kg as a subcutaneous injection every 3 weeks with a 3 week prednisone boost of 1 mg/kg/day (max 60 mg) to be completed in 3 patients without untoward events
- Sotatercept Cohort 5b: Cohort 5b: Sotatercept 1 mg/kg given as a subcutaneous injection every 3 weeks - to be completed in 3 patients without untoward events
Period: Overall Study
Arm/Group | Sotatercept Cohort 1 | Sotatercept Cohort 2 | Sotatercept Cohort 3 | Sotatercept With Prednisone Boost Cohort 4a | Sotatercept Cohort 4b | Sotatercept With Prednisone Boost Cohort 5a | Sotatercept Cohort 5b
Started | 3 | 4 | 4 | 2 | 3 | 0 | 3
Completed | 3 | 2 | 2 | 2 | 3 | 0 | 1
Not Completed | 0 | 2 | 2 | 0 | 0 | 0 | 2
Not completed — Screen failure | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: There were no subjects in Cohort 5a at the time of the closure of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotatercept Cohort 1 | Sotatercept Cohort 2 | Sotatercept Cohort 3 | Sotatercept With Prednisone Boost Cohort 4a | Sotatercept Cohort 4b | Sotatercept With Prednisone Boost Cohort 5a | Sotatercept Cohort 5b | Total
Number analyzed (Participants) | 3 | 4 | 4 | 2 | 3 | 0 | 3 | 19
Age, Continuous [Median (Full Range); unit: years] — Population: Three subjects of the original consented subjects did not meet the eligibility criteria and were screen failures. Three subjects met the criteria for enrollment but did not complete the study to be analyzed as the subjects were terminated early.
  years
    number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 0 | 1 | 13
    (all) | 36 [25 to 41] | 34 [27 to 42] | 32 [20 to 43] | 39 [31 to 47] | 31 [20 to 36] |  | 37 [37 to 37] | 35 [20 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three subjects of the original consented subjects did not meet the eligibility criteria and were screen failures. Three subjects met the criteria for enrollment but did not complete the study to be analyzed as the subjects were terminated early.
  Participants
    number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 0 | 1 | 13
    Female | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 5
    Male | 3 | 0 | 1 | 1 | 2 | 0 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three subjects of the original consented subjects did not meet the eligibility criteria and were screen failures. Three subjects met the criteria for enrollment but did not complete the study to be analyzed as the subjects were terminated early.
  Participants
    number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 0 | 1 | 13
    Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3
    Not Hispanic or Latino | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 10
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 1 | 2 | 2 | 0 | 3 | 13
  More than one race | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response and Partial Response
Description: Complete response is transfusion independence with hemoglobin >9 gm/dl; partial response is transfusion dependence with hemoglobin < 9gm/dl with an increase in reticulocyte count over baseline
Time Frame: 9 months
Population: Only subjects who completed the trial are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept Cohort 1 | Sotatercept Cohort 2 | Sotatercept Cohort 3 | Sotatercept With Prednisone Boost Cohort 4a | Sotatercept Cohort 4b | Sotatercept With Prednisone Boost Cohort 5a | Sotatercept Cohort 5b
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 0 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Severe Adverse Events Attributable to Study Drug
Description: Assess severity of adverse events and relationship to sotatercept according to the currently active minor version of the NCI Common Terminology for Adverse Events version 4.0
Time Frame: 9 months
Population: Only subjects who completed the trial are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept Cohort 1 | Sotatercept Cohort 2 | Sotatercept Cohort 3 | Sotatercept With Prednisone Boost Cohort 4a | Sotatercept Cohort 4b | Sotatercept With Prednisone Boost Cohort 5a | Sotatercept Cohort 5b
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 0 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the time the subject was on study, a total of 9 months.
Description: Cohort 5a had no subjects enrolled.
Arm/Group | Sotatercept Cohort 1 | Sotatercept Cohort 2 | Sotatercept Cohort 3 | Sotatercept With Prednisone Boost Cohort 4a | Sotatercept Cohort 4b | Sotatercept With Prednisone Boost Cohort 5a | Sotatercept Cohort 5b
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/2 | 0/3 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/2 | 0/2 | 0/2 | 1/3 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/2 | 0/3 | 0/0 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept Cohort 1 (N=3) | Sotatercept Cohort 2 (N=2) | Sotatercept Cohort 3 (N=2) | Sotatercept With Prednisone Boost Cohort 4a (N=2) | Sotatercept Cohort 4b (N=3) | Sotatercept With Prednisone Boost Cohort 5a (N=0) | Sotatercept Cohort 5b (N=1)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Cellulitis at injection site of non-study drug with episode of neutropenia.
Hospitalization (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Shortness of breath and fatigue noted with hypothyroidism
Elevated liver function tests (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject with elevated LFTs found to have EBV infection .

LIMITATIONS AND CAVEATS:
Early termination of 3 subjects lead to small numbers of subjects analyzed, as does the early closure of the study.

Time to response was unable to be evaluated as no subjects attained response. Response duration was also not evaluated as no subjects responded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT01464164/Prot_SAP_000.pdf